CLINICAL TRIAL: NCT04101994
Title: Augmented Effects of Virtual-reality Cycling Training on Upper Limb Motor Functions by Noninvasive Brain Stimulation in Patients With Cerebral Palsy
Brief Title: Augmented Effects of Virtual-reality Cycling Training on Upper Limb Motor Functions by NIBS in Patients With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201701518A0
Record Dates: First submitted 2019-09-22; First posted 2019-09-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: virtual cycling training; Non-invasive brain stimulation; repetitive transcranial magnetic stimulation; transcranial electric stimulation
MeSH Terms: conditions — Cerebral Palsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- VCT and real rTMS (Experimental): In virtual cycling training and intermittent theta burst stimulation group (VCT + iTBS group), they received VCT and iTBS (80% of active motor threshold) on affected hemisphere.
  Interventions: Device: Virtual cycling training; Device: Repetitive transcranial magnetic stimulation
- VCT and sham rTMS (Experimental): In virtual cycling training and sham theta burst stimulation group (VCT + iTBS group), they received VCT and sham TBS stimulation.
  Interventions: Device: Virtual cycling training; Device: Repetitive transcranial magnetic stimulation
- real rTMS (Experimental): In intermittent theta burst stimulation (iTBS group), they received iTBS (80% of active motor threshold) on affected hemisphere.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- sham rTMS (Sham Comparator): In sham theta burst stimulation (sham TBS group), they received sham TBS stimulation.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- VCT and real TES (Experimental): In virtual cycling training and transcranial electric stimulation group (VCT + TES group), they received TES stimulation over motor cortex.
  Interventions: Device: Virtual cycling training; Device: Transcranial electric stimulation
- VCT and sham TES (Experimental): In virtual cycling training and sham transcranial electric stimulation group (VCT + sham TES group), they received VCT and sham TES stimulation.
  Interventions: Device: Virtual cycling training; Device: Transcranial electric stimulation
- real TES (Experimental): In transcranial electric stimulation group (TES group), they received TES stimulation over motor cortex.
  Interventions: Device: Transcranial electric stimulation
- sham TES (Sham Comparator): In sham transcranial electric stimulation group (sham TES group), they received sham TES stimulation.
  Interventions: Device: Transcranial electric stimulation

INTERVENTIONS:
Device: Virtual cycling training — Virtual cycling training is a convenient and easy approach for muscle strengthening.
  Arms: VCT and real TES; VCT and real rTMS; VCT and sham TES; VCT and sham rTMS
Device: Repetitive transcranial magnetic stimulation — Intermittent theta burst stimulation produces short TBS trains intermittently to facilitate cortical excitability.
  Arms: VCT and real rTMS; VCT and sham rTMS; real rTMS; sham rTMS
Device: Transcranial electric stimulation — TES is a constant current with low intensity delivered to the skull through surface electrodes.
  Arms: VCT and real TES; VCT and sham TES; real TES; sham TES

SUMMARY:
Cerebral palsy (CP) is the most common childhood motor disability. Weakness, spasticity, and loss of dexterity are the major problems in patients with CP. A novel virtual-reality cycling training (VCT) program was to enhance promising muscle strength and motor function through promoting the participant compliance and motivation. Non-invasive brain stimulation (NIBS), such as repetitive transcranial magnetic stimulation (rTMS) and transcranial electric stimulation (TES) has potential to augment the training effects in motor neurorehabilitation via the modulation on neuroplasticity. Therefore, this study propose a novel intervention protocol to induce superior benefits on upper extremity (UE) motor function in patients with CP.

DETAILED DESCRIPTION:
This study aims to investigate the augmented effects of VCT on neuromotor control and UE motor function by NIBS in patients with CP. We hypothesize that NIBS can augment the VCT effects on neuromotor control and UE motor function in patients with CP because combined therapy integrated peripheral modification techniques (VCT) and central modulation (NIBS). These effects may further enhance the activity of daily living (ADL), participation, and health related quality of life (HRQOL). This project is executed in the following two phases: to investigate the augmented effects of VCT on neuromotor control and UE motor function in patients with CP by rTMS in phase 1 (0-1.5 years) and tCS in phase 2 (1.5-3 years).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CP according to clinical criteria
* Age 5-20 years
* No use of botulinum toxin in the past 4 months
* No significant perceptual or communication disturbances
* No other peripheral or central nervous system dysfunction
* No active inflammatory or pathologic changes in upper limb joints during the previous 6 months
* No active medical problems, such as pneumonia, upper gastrointestinal bleeding, or urinary tract infection
* No active problems of epilepsy and EEG without epileptiform discharge

Exclusion Criteria:

* Metabolic disorders, such as inborn error of metabolism, electrolyte, and endocrine disorders
* Active infectious disease, such as meningitis and encephalitis
* Patients with active medical problems, such as pneumonia, upper gastrointestinal bleeding, or urinary tract infection
* Poor compliance or intolerance for the TMS therapy
* Subjects with metallic implants or pregnancy.
* EEG show epileptiform discharge
* Patients with family history of epilipsy
* Patients with symptoms that are restricted from tDCS, such as epilepsy, migraine and unstable health condition

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Bruininks- Oseretsky Test of Motor Proficiency II at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The Bruininks- Oseretsky Test of Motor Proficiency II (BOT-2) provides an overview of fine and gross motor skills in children and school-aged adolescents.
Change from baseline Goal Attainment Scale at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  Goal Attainment Scale (GAS) is used to help a person with cerebral palsy and their family develop personal goals for therapy (for each item minimum value is -2 and maximum value is 2, higher scores mean a better outcome).

SECONDARY OUTCOMES:
Change from baseline Melbourne Assessment 2 at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The Melbourne Assessment 2 (MA2) is a valid and reliable tool for evaluating quality of upper limb movement in children with a neurological impairment aged 2.5 to 15 years.
Change from baseline Quality of upper extremity skills test at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The Quality of upper extremity skills test (QUEST) is an outcome measure that evaluates movement patterns and hand function in children with cerebral palsy.
Change from baseline Box and block test at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The Box and Block Test (BBT) measures unilateral gross manual dexterity.
Change from baseline Nine-Hole test at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The Nine-Hole Peg Test (NHPT) is used to measure finger dexterity in patients with various neurological diagnoses.
Change from baseline Functional Independence Measure at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  Functional Independence Measure for Children:Applicable to infants and adolescents. The main purpose is to understand and track children's life function performance, progress and goal achievement. There are three main areas: self-care, mobility, and cognition. The score is from 1 to 7 points, 1 is completely dependent, and 7 is completely independent.
Change from baseline Pediatric Motor Activity Log at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The Pediatric Motor Activity Log (PMAL) is a structured interview intended to examine how often and how well a child uses his/her involved upper extremity (UE) in their natural environment outside the therapeutic setting.
Change from baseline ABILHAND Questionnaire at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The ABILHAND questionnaire assesses bimanual ability as an interview-based test focused on the patient's perceived difficulty. The ABILHAND-KIDS questionnaire is filled in by the parent of the child by rating the child's perceived difficulty of bimanual activities.
Change from baseline Assessment of Preschool Children's Participation at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  Preferences for Activity of Children(APCP): For children between the ages of two and five, the questionnaire model is used to allow parents to circle the level. There are 45 questions in total, so that the case or parent can review the activities in the past 4 months and ask if the child have done this activity (1 point means yes, 0 points means no).
Change from baseline Children Assessment of Participation and Enjoyment at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  Children Assessment of Participation and Enjoyment(CAPE): Applicable to children or adolescents between the ages of six and twenty one, through questionnaires through self-reports or interviews, a total of 55 questions, asking children about the activities involved in the past four months (1 point for yes, 0 for no).
Change from baseline Cerebral Palsy Quality of Life at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The comparison of baseline of Cerebral Palsy Quality of Life for CP after different therapy.
Change from baseline Motor Evoked Potential at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The comparison of baseline of Motor Evoked Potential for CP after different therapy.
Change from baseline Myoton at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The comparison of baseline of Myoton for CP after different therapy.
Change from baseline Hand dynamometer at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  The comparison of baseline of hand dynamometer for CP after different therapy.
Change from baseline Motion analysis at after six weeks of treatment and three month | baseline, after 6 weeks of treatment, 3 months
  All participants will be instructed to perform a series of upper-extremity tasks. The tasks include reaching and grasping. An 8-camera motion analysis system (Vicon system, 3-D Oxfort Metrics Ltd, Oxford, UK) is used in conjunction with a personal computer to capture the movement of markers placed on the participant's body; analog signals were collected simultaneously. Movements were recorded at 120 Hz and digitally low-pass filtered at 5 Hz using a second-order Butterworth filter. Reference markers are placed on the distal interphalangeal joints of the thumb and index finger, the styloid process of the ulna, proximal end of the second metacarpal, and the object.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD, PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No